CLINICAL TRIAL: NCT00943618
Title: Effectiveness of Varenicline vs. Varenicline Plus Bupropion or Placebo for Smoking Cessation
Brief Title: Combining Varenicline and Bupropion for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-0850; R01DA024709-01A1 (NIH); NCI-2011-01101 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Nicotine Withdrawal; Smoking Reduction; Varenicline; Chantix; Bupropion; Zyban
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction | interventions — Varenicline; Bupropion; Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Varenicline and Bupropion
  Interventions: Drug: Varenicline; Drug: Bupropion; Behavioral: Counseling/Phone Calls
- Group 2 (Placebo Comparator): Varenicline and Placebo
  Interventions: Drug: Varenicline; Other: Placebo; Behavioral: Counseling/Phone Calls
- Group 3 (Placebo Comparator): Placebo that looks like varenicline and a placebo that looks like bupropion.
  Interventions: Other: Placebo; Behavioral: Counseling/Phone Calls

INTERVENTIONS:
Drug: Varenicline — On Days 1-3, .5mg tablet by mouth in the morning. Beginning on Day 4, and then every day after that, .5mg tablet by mouth in the morning and .5mg tablet by mouth in the evening (for a total of 2 doses).
  Other Names: Chantix
  Arms: Group 1; Group 2
Drug: Bupropion — On Days 1-3, 150 mg tablet by mouth in the morning. Beginning on Day 4, and then every day after that, 150 mg tablet by mouth in the morning and 150 mg tablet by mouth in the evening (for a total of 2 doses).
  Other Names: Zyban
  Arms: Group 1
Other: Placebo — On Days 1-3, 1 tablet by mouth of placebo that looks like the study drug in the morning. Beginning on Day 4, and then every day after that, 1 tablet by mouth in the morning and 1 tablet by mouth in the evening for a total of 2 doses of the placebo each day.
  Arms: Group 2; Group 3
Behavioral: Counseling/Phone Calls — Brief-behavioral counseling sessions (10-15 minutes) provided to all participants once per week for 12 weeks. One support phone call conducted 3 days after the target quit date.

SUMMARY:
The goal of this clinical research study is learn if the combination of Chantix (varenicline) and Zyban (bupropion) is more effective at helping people to quit smoking than varenicline when given alone. Researchers also want to learn if this drug combination can reduce cravings and other negative symptoms of nicotine withdrawal better than varenicline does alone. The safety of this drug combination will also be tested.

DETAILED DESCRIPTION:
The Study Drugs:

Bupropion and varenicline are designed to imitate the effects that nicotine has on the body. This may reduce cigarette cravings and help patients quit smoking.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of a dice) to 1 of 3 treatment groups.

* If you are in Group 1, you will receive varenicline and bupropion.
* If you are in Group 2, you will receive varenicline and a placebo. A placebo is a substance that looks like the study drug (in this case, bupropion) but that has no active ingredients.
* If you are in Group 3, you will receive a placebo that looks like varenicline and a placebo that looks like bupropion.

You will have a higher chance (5 out of 6) of receiving study drug than receiving just placebo. Equal numbers of patients will be in Groups 1 and 2. Neither you nor the study doctor will know to which group you are assigned. However, if needed for your safety, the study staff will be able to find out which study drug you are receiving.

Study Drug Administration:

You will begin taking the study drugs/placebo 1 to 10 days after the first study visit. A dose of the study drug/placebo combination will be made up of 1 tablet of varenicline or placebo and 1 tablet of bupropion or placebo. You should take each dose of study drugs/placebo with a cup (8 oz.) of water after eating a full meal.

On Days 1-3, you will take 1 dose of the study drug/placebo combination in the morning.

Beginning on Day 4, and then every day after that, you will take 1 dose in the morning and 1 dose in the evening (for a total of 2 doses of the study drug/placebo combination each day). You must return any study drug bottles as well as any unused study drug to a study staff member at each study visit.

You will be given a smoking diary to record how many cigarettes you smoke (if any) each day while you are on study. You must turn in this diary at each study visit.

Study Visits:

About 1 time each week while you are taking the study drugs/placebo, the following tests and procedures will be performed:

* Your weight and blood pressure will be measured.
* Your CO level will be measured.
* You will be asked about any other drugs you may be taking and about any side effects you may be having.
* You will answer 8 questionnaires about several topics, including depression, suicide, your smoking behavior, any effects from the study drugs, and any symptoms of attention-deficit hyperactivity disorder (ADHD). These should take about 30-45 minutes total to complete.
* You will do tasks that will measure your logic and attention. These will take about 15 -20 minutes to complete.
* You will receive counseling about quitting smoking in which you discuss possible "triggers" for smoking and strategies for dealing with quitting smoking. These sessions will take about 15 minutes each time.

During counseling at the first study visit, you will set a "quit date" for stopping smoking for about 1 week after you start taking the study drug. You should not quit smoking before the quit date. You should stay smoke-free after the quit date. Additionally, you will be given a medication instruction sheet, a card with emergency contact information, and a participant manual to help you follow along with the topics discussed during counseling.

At Week 2, saliva will be collected to check your cotinine level.

At Week 4, blood (about 2 teaspoons) will be drawn to assess liver and kidney function.

Lab Sessions:

You may be asked to take part in lab sessions during Visits 1, 2, and 6 to test your brain activity and attention span. You will be asked to watch slides and listen to a series of tones. The slides will include pictures of people, nature, and artwork. Slides showing nude people, medical procedures, and victims of car crashes will also be shown. You will be shown examples of these slides before beginning the procedure and given the opportunity to withdraw from the study.

During the lab sessions, your brain electrical activity (EEG) will be monitored. To do this, small sensors will be placed on your scalp and face. You should not drink more than 2 cups of coffee or other caffeinated drinks for at least 2.5 hours before each session. At the first lab session, you may be asked to smoke a cigarette if the doctor thinks it is needed for you to exhibit your normal smoking behavior.

Length of Study:

You will receive the study drug for up to 12 weeks. However, the entire length of the study is about 13 months (55 weeks), which includes 3, 6, and 12-month post-quit follow up visits. You will be taken off study if the doctor thinks it is in your best interest.

End-of-Study Visit:

After you have finished taking the study drugs/placebo, the following tests and procedures will be performed:

* Your weight and blood pressure will be measured.
* Your CO level will be measured.
* You will be asked about any side effects you may be having and about any other drugs you may be taking.
* Blood (about 2 teaspoons) will be drawn to assess liver and kidney function.
* You will answer the same questionnaires you completed at the regular study visits. These should take about 30-45 minutes total to complete.
* Saliva will be collected to measure your cotinine level.

Follow-Up Visits:

About 3, 6, and 12 months after you have stopped smoking, the following tests and procedures will be performed:

* Your weight, heart rate, and blood pressure will be measured.
* Your CO level will be measured.
* You will be asked about any side effects you may be having and about any other drugs you may be taking.
* You will answer the same questionnaires you completed at the regular study visits. These should take about 30-45 minutes total to complete.
* Saliva will be collected to measure your cotinine level.

You will be called by the study staff 1 day before your quit date, 3 days after your quit date, and at Weeks 14, 20, 34, 42, and 48 weeks after your quit date to check on your progress in quitting smoking. Each call should take about 10-15 minutes.

This is an investigational study. Varenicline and bupropion are both FDA approved and commercially available to help people stop smoking. The use of the drugs in combination is investigational.

Up to 385 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25-70 years old
2. Smoking 5 or more cigarettes per day, on average, within the 2 months preceding the screening visit and expired CO of greater than or equal to 6ppm.
3. Able to follow verbal and written instructions in English and complete all aspects of the study
4. Provide informed consent and agree to all assessments and study procedures
5. Have an address and home telephone number where they may be reached
6. Be the only participant in their household

Exclusion Criteria:

1. Within the month immediately preceding the screening visit, use of any form of tobacco products other than cigarettes on 3 or more days within a week if the individual refuses to refrain from such tobacco use during the course of the study.
2. Within the month immediately preceding the screening visit, use of marijuana in any form on 3 or more days within a week
3. Within the two weeks immediately preceding the screening visit, involvement on more than 3 days in any formal smoking cessation activities
4. Treatment on a continuous basis within 2 weeks before the screening visit: any contraindicated medication for Varenicline or Bupropion. Classes of contraindicated medications include, but are not limited to, antiasthmatics, antipsychotics, some antidepressants, antihypertensives, antiarrhythmics, antineoplastics, some antiseizures, and MAO inhibitors (See Appendix U for specific list of excluded and precautionary medications).
5. Uncontrolled hypertension (average reading of systolic blood pressure greater than 150 or diastolic blood pressure greater than 95) or other major contraindications for Bupropion or Varenicline (See section on Screening).
6. Severe renal impairment (Creatinine Clearance less than 30 ml/min/1.73 m2).
7. Laboratory evaluations outside normal limits and of potential clinical significance in the opinion of the investigator.
8. Meet current criteria for psychiatric disorders or substance abuse as assessed by the MINI plus (major depressive episode) and the MINI for items B, D, I, J (Alcohol Addendum-past 6 months only), K, L, M and N including a past manic or hypomanic episode as well as a lifetime psychotic disorder.
9. Individuals rated as moderate (6 - 9) to high (10 or greater) on suicidality as assessed by Module C of the MINI.
10. Psychiatric hospitalization within 1 year of screening date.
11. A positive urine pregnancy test during the screening period. Women who are two years post menopausal, or who have had a tubal ligation or a partial or full hysterectomy will not be subject to a urine pregnancy test.
12. Pregnant, breast-feeding or of childbearing potential and is not protected by a medically acceptable, effective method of birth control while enrolled in the study. Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD). Contraceptive measures sold for emergency use after unprotected sex, are not acceptable methods for routine use.
13. Use of Varenicline or Bupropion within two weeks before the screening visit.
14. History of hypersensitivity or allergic reaction to Varenicline, tricyclic antidepressant, Bupropion (Wellbutrin, Zyban) or similar chemical classes or any component of these formulations.
15. Current or previous history of a seizure disorder.
16. Current or previous history of anorexia.
17. Subject considered by the investigator as unsuitable candidate for receipt of an investigational drug or unstable to be followed up throughout the entire duration of the study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Cinciripini, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Cinciripini PM, Minnix JA, Green CE, Robinson JD, Engelmann JM, Versace F, Wetter DW, Shete S, Karam-Hage M. An RCT with the combination of varenicline and bupropion for smoking cessation: clinical implications for front line use. Addiction. 2018 Apr 21:10.1111/add.14250. doi: 10.1111/add.14250. Online ahead of print. PMID 29679432
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Paid and unpaid media advertising from May 2010 to July 2013 recruited volunteer smokers from the Houston, Texas metropolitan area. Inclusion criteria included: 25- 65 years of age; smoke five or more cigarettes per day (CPD); baseline expired carbon monoxide (CO) level greater than 6 parts per million (p.m.); fluent in English; stable residency.
Pre-assignment Details: 641 patients were consented to this study; 250 patients were screen failures.
Groups:
- Varenicline + Bupropion: Smokers in varenicline + bupropion took 0.5 mg varenicline once per day for the first three days and 0.5 mg bid (am and pm) for the next 4 days. They also took 150 mg bupropion (SR once per day for the first 3 days followed by 150mg bid for the next 4 days. From week 2-12 smokers in the VB group will take 1mg of varenicline and one active 150 mg bupropion tablet twice per day.
- Varenicline: Smokers in varenicline group took took 0.5 mg varenicline once per day for the first three days and 0.5 mg bid (am and pm) for the next 4 days. They also took a matching bupropion placebo on the same schedule as those in the varenicline + bupropion group. From week 2-12, smokers in the varenicline group took 1mg of varenicline and one bupropion matching placebo twice per day.
- Placebo: Smokers in the placebo group took a matching varenicline and bupropion placebos on the same schedule as the varenicline group took varenicline and the bupropion group took bupropion, respectively.
Period: Overall Study
Arm/Group | Varenicline + Bupropion | Varenicline | Placebo
Started | 163 | 166 | 56
Completed | 108 | 89 | 25
Not Completed | 55 | 77 | 31
Not completed — Lost to Follow-up | 38 | 48 | 20
Not completed — Discontinued Medication | 17 | 29 | 11

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated participants, i.e. Intention to Treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline + Bupropion | Varenicline | Placebo | Total
Number analyzed (Participants) | 163 | 166 | 56 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.36 (9.38) | 48.75 (10.89) | 48.48 (10.33) | 48.97 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 68 | 24 | 160
  Male | 95 | 98 | 32 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 6 | 30
  Not Hispanic or Latino | 146 | 146 | 48 | 340
  Unknown or Not Reported | 7 | 6 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 5 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 44 | 43 | 16 | 103
  White | 106 | 110 | 36 | 252
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 8 | 5 | 1 | 14
Region of Enrollment [Number; unit: participants]
  United States | 163 | 166 | 56 | 385
Marital Status [Number; unit: percentage of participants]
  Married or Living with partner | 42.94 | 53.01 | 62.50 | 50.13
  Other | 57.06 | 46.99 | 37.50 | 49.87
Employment Status [Number; unit: percentage of participants]
  Employed/Student | 82.72 | 80.72 | 78.57 | 81.25
  Unemployed | 17.28 | 19.28 | 21.43 | 18.75
Depression History [Count of Participants; unit: Participants] — Depression history indicates whether the participant had a history of depression (positive) or did not have a history of depression (negative). It is a proportions/percentages characteristic.
  Participants
    Positive | 9 | 10 | 4 | 23
    Negative | 154 | 156 | 52 | 362
Years of education [Mean (Standard Deviation); unit: years] | 13.89 (2.11) | 13.60 (1.92) | 13.80 (1.89) | 13.75 (2)
Current Smoking Rate [Mean (Standard Deviation); unit: cigs per day] | 19.64 (9.49) | 19.02 (9.49) | 19.71 (11.20) | 19.66 (9.45)
Number of Previous Quit Attempts [Mean (Standard Deviation); unit: Number of quit attempts] | 7.58 (13.51) | 5.83 (9.22) | 6.12 (13.90) | 6.62 (11.94)
Age started smoking [Mean (Standard Deviation); unit: years] | 18.41 (5.15) | 18.16 (60.16) | 16.48 (3.43) | 18.02 (5.44)
Fagerström Test for Nicotine Dependence (FTND) Total Score [Mean (Standard Deviation); unit: score on a scale] — FTND (Fagerström Test for Nicotine Dependence) SCORE (Range = 0-10) Higher scores indicate more dependence.
  score on a scale | 4.74 (2.01) | 4.65 (2.04) | 5.34 (2.24) | 4.79 (2.07)
Center for Epidemiologic Studies Depression Scale (CESD) [Mean (Standard Deviation); unit: score on a scale] — CESD consists of twenty items that are rated on a four-point likert scale (from 1: rarely or none of the time to 4: most or all of the time). Scores range from zero to sixty. Higher scores indicated a higher frequency of depressive symptoms. CORE (Range = 0-60). Higher scores indicate more depression.
  score on a scale | 5.82 (5.37) | 7.76 (7.07) | 6.59 (6.17) | 6.73 (6.27)
Positive and Negative Affect Schedule (PANAS) [Mean (Standard Deviation); unit: units on a scale] — The questionnaire contains 20 items on two subscales that assess a person's positive and negative trait affect using a 5-point scale (1= "very slightly or not at all"; 5=" extremely"). SCORE (Range 10-50). Higher scores in the PANAS Negative scale indicate higher negative emotions". "Higher scores in the PANAS Positive scale indicate higher positive emotions
  units on a scale
    PANAS Negative | 14.56 (4.93) | 14.93 (5.31) | 14.44 (4.39) | 14.70 (5.02)
    PANAS Positive | 34.08 (7.64) | 33.26 (7.43) | 33.84 (8.80) | 33.69 (7.72)
Wisconsin Smoking Withdrawal Scale (WSWS) [Mean (Standard Deviation); unit: score on a scale] — Wisconsin Withdrawal Scale (WSWS) contains 7 factors: Anger, Anxiety, Sadness, Concentration, Craving, Sleep, and Hunger. The items are scored on a 5-point Likert type scale (0 = strongly disagree, 4 = strongly agree). SCORE (Range= 0-12). Higher scores in the Anger, Anxiety, Sadness, Craving and Hunger scale indicate worse outcome; higher scores in the Concentration indicates lack of concentration, higher score in sleep scale indicate more problems sleeping.
  score on a scale
    Anger | 3.57 (2.25) | 4.01 (2.48) | 3.67 (23.8) | 3.77 (2.37)
    Anxiety | 6.80 (2.74) | 6.96 (2.99) | 7.15 (2.76) | 6.92 (2.84)
    Concentration | 3.80 (2.05) | 3.84 (2.02) | 3.69 (1.99) | 3.80 (2.02)
    Craving | 9.40 (2.63) | 9.86 (2.94) | 9.87 (2.85) | 9.67 (2.80)
    Hunger | 9.67 (3.39) | 10.46 (3.50) | 10.31 (3.44) | 10.10 (3.46)
    Sadness | 4.38 (2.21) | 4.76 (2.48) | 4.55 (2.04) | 4.57 (2.31)
    Sleep | 7.91 (4.04) | 8.52 (4.48) | 8.16 (4.47) | 8.21 (4.29)
Wisconsin Index of Smoking Dependence Motives (WISDM) [Mean (Standard Deviation); unit: units on a scale] — (WISDM) is comprised of 68 items designed to assess 13 different motivational domains: affiliative attachment, automaticity, loss of control, behavioral choice/melioration, cognitive enhancement, craving, cue exposure/associative processes, negative reinforcement, positive reinforcement, social/environmental goads, taste/sensory properties, tolerance, and weight control. The WISDM consists of 68 items that are rated on a 7-point Likert scale. SCORE (Range = 1-7). Subscales are summed to provide a total score (Range = 11-77). In all cases higher scores indicate worse outcomes.
  units on a scale
    WISDM-Affect | 4.83 (2.00) | 4.75 (2.01) | 5.22 (1.97) | 4.85 (2.00)
    WISDM-Affiliation | 4.20 (2.13) | 3.87 (2.22) | 4.41 (2.42) | 4.09 (2.22)
    WISDM-Automaticity | 6.05 (2.02) | 5.57 (2.17) | 6.42 (2.11) | 5.90 (2.11)
    WISDM-Cognitive | 4.66 (2.09) | 4.37 (2.17) | 4.82 (2.05) | 4.56 (2.12)
    WISDM-Control | 6.17 (1.73) | 6.32 (1.87) | 6.51 (2.09) | 6.28 (1.85)
    WISDM-Craving | 6.11 (1.62) | 5.95 (1.78) | 6.53 (1.83) | 6.11 (1.73)
    WISDM-Cue Exposure-Associative Processes | 5.36 (1.82) | 5.34 (2.02) | 5.56 (1.74) | 5.38 (1.90)
    WISDM-Social-Environmental Goads | 4.00 (2.22) | 3.77 (2.54) | 4.25 (2.59) | 3.94 (2.42)
    WISDM-Primary Dependence Motives | 6.08 (1.53) | 5.96 (1.64) | 6.43 (1.75) | 6.08 (1.61)
    WISDM-Secondary Dependence Motives | 4.57 (1.36) | 4.38 (1.48) | 4.71 (1.46) | 4.51 (1.43)
    WISDM-Taste and Sensory Processes | 5.52 (2.06) | 5.29 (2.27) | 5.50 (2.11) | 5.41 (2.16)
    WISDM-Tolerance | 6.01 (2.04) | 6.01 (2.11) | 6.26 (2.04) | 6.04 (2.07)
    WISDM-Weight Control | 3.40 (1.93) | 3.29 (2.10) | 3.18 (2.12) | 3.32 (2.03)
    WISDM-Total | 56.32 (14.11) | 54.54 (15.66) | 58.65 (15.53) | 55.89 (15.03)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence at 12 Months
Description: Prolonged Abstinence is defined as no smoking from the quit date to 12 Months post quit date.
Time Frame: From quit date to 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Bupropion | Varenicline | Placebo
Number analyzed (Participants) | 163 | 166 | 56
Participants | 30 | 33 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Varenicline + Bupropion | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/166 | 0/56
Serious Adverse Events (participants affected / at risk) | 8/163 | 4/166 | 1/56
Other Adverse Events (participants affected / at risk) | 160/163 | 156/166 | 50/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline + Bupropion (N=163) | Varenicline (N=166) | Placebo (N=56)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Chest pain-cardiac (Cardiac disorders) | 0 | 0 | 1
Cholecystitis (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Delerium (Psychiatric disorders) | 1 | 0 | 0
Depressive Symptoms (Psychiatric disorders) | 1 | 0 | 0
Disturbance in attention (Psychiatric disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Flashing lights (Eye disorders) | 1 | 0 | 0
Floaters (Eye disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Infection and infestation - Strep Throat (Infections and infestations) | 0 | 2 | 0
Infection and infestation - Tonsillitis (Infections and infestations) | 0 | 1 | 0
Influenza (General disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Reproductive system and breast disorders-other: uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia/Palpitations (Cardiac disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline + Bupropion (N=163) | Varenicline (N=166) | Placebo (N=56)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 4 | 4 | 2
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Tachycardia/Palpitations (Cardiac disorders) | 3 | 7 | 2
Earache (Ear and labyrinth disorders) | 0 | 1 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 6 | 1 | 0
Endocrine disorders, other-excessive thirst (Endocrine disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 8 | 5 | 2
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Eye irritation (Eye disorders) | 4 | 12 | 3
Flashing lights (Eye disorders) | 1 | 0 | 0
Floaters (General disorders) | 1 | 0 | 0
Photosensitivity (Eye disorders) | 0 | 1 | 0
eye disorders, other-eye twitching (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 22 | 16 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Blood in Stool (Gastrointestinal disorders) | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 4 | 5 | 1
Cecal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 22 | 19 | 3
Diverticulitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 21 | 2
Dry mouth (Gastrointestinal disorders) | 28 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 11 | 11 | 4
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 12 | 10 | 4
Gallbladder obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastro-esophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0
Gastrointestinal anastomotic leak (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 2 | 1
Gastrointestinal disorders, other-softer stools (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorders, other-increased salivation (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hiccups (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 47 | 64 | 7
Oral pain (Gastrointestinal disorders) | 2 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 7 | 7 | 3
Vomiting (Gastrointestinal disorders) | 17 | 18 | 2
Appetite, decreased (Gastrointestinal disorders) | 20 | 9 | 0
Appetite, increased (Gastrointestinal disorders) | 24 | 29 | 5
Chest Pain - non cardiac (General disorders) | 4 | 9 | 1
Dehydration (General disorders) | 1 | 5 | 1
Dizziness (General disorders) | 29 | 31 | 10
Face Edema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 22 | 22 | 7
General Disorders and administration site conditions - Other, Hyperthermia (General disorders) | 1 | 0 | 0
General disorders and administration site conditions, other -blood from throat (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, feeling speedy (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0 | 0
Influenza (General disorders) | 28 | 25 | 11
Vertigo (General disorders) | 2 | 1 | 0
Weight gain (General disorders) | 18 | 28 | 3
Weight loss (General disorders) | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Allergy, Seasonal (Immune system disorders) | 1 | 0 | 0
Immune system disorders - Shingles (Immune system disorders) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 5 | 3 | 0
Gum infection (Infections and infestations) | 1 | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 2
Infection and infestation - Other - swollen lymph nodes (Infections and infestations) | 0 | 1 | 0
Infection and infestation - Strep Throat (Infections and infestations) | 0 | 1 | 0
Infection and infestation - Tonsillitis (Infections and infestations) | 0 | 1 | 0
Infections & infestations, other-mycobacterium avium complex) (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1
Infections and infestations, other-fever blisters (Infections and infestations) | 1 | 1 | 0
Infections and infestations, other-infection of R hand (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Mucositis oral (Infections and infestations) | 1 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis - bacterial (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 4 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 9 | 11 | 4
Alanine aminotransferase increased (General disorders) | 12 | 12 | 1
Aspartate aminotransferase increased (General disorders) | 11 | 15 | 2
Bilirubin Increased (General disorders) | 2 | 0 | 0
Blood Bilirubin Increased (General disorders) | 0 | 1 | 0
Creatinine increased (General disorders) | 17 | 1 | 1
GGT increased (General disorders) | 16 | 10 | 1
Hepatobiliary disorders - Elevated GGT (General disorders) | 0 | 1 | 0
Investigations - Increased Alcohol Consumption (General disorders) | 1 | 0 | 0
Investigations, Other - Specify (General disorders) | 0 | 1 | 0
Investigations-other (abnormal EKG) (Investigations) | 0 | 0 | 1
Vascular disorders, other-hypercholesterolemia (General disorders) | 1 | 0 | 0
General disorders & administration site conditions - Diaphoresis (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 7 | 2 | 1
Metabolism and nutrition disorders, other-low B12 levels (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Edema (Musculoskeletal and connective tissue disorders) | 16 | 5 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Inflammation Gluteus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Localized edema (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 45 | 50 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 4 | 1
PERIPHERAL EDEMA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasms benign, malignant, and unspecified (incl cysts & polyps) - other uterine fibroids (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasms, benign, malignant, & unspecified, (incl cysts & polyps) other-spot on cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 29 | 31 | 10
Dysgeusia (Nervous system disorders) | 20 | 6 | 2
FALL (Nervous system disorders) | 1 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 33 | 35 | 14
Nervous System disorders, other - Somniloquy (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder other-jittery (Nervous system disorders) | 2 | 0 | 0
Nervous system disorder, other-feeling heart beating (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder, other-headrushes (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders, other-Migraine (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders, other-lightheadedness (Nervous system disorders) | 0 | 2 | 0
Neurology - other (Nervous system disorders) | 0 | 1 | 0
Olfactory nerve disorder (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0
Sensory disturbance (Nervous system disorders) | 11 | 12 | 1
Slurred Speech (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 4 | 2 | 1
Asthenia (Psychiatric disorders) | 0 | 1 | 0
Abnormal Dreams (Psychiatric disorders) | 42 | 57 | 6
Anxiety symptoms (Psychiatric disorders) | 38 | 26 | 10
Depressive Symptoms (Psychiatric disorders) | 39 | 40 | 14
Disturbance in attention (Psychiatric disorders) | 31 | 27 | 10
Hallucinations (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 87 | 60 | 17
Irritability (Psychiatric disorders) | 32 | 42 | 10
Personality change (Psychiatric disorders) | 3 | 3 | 0
Psychiatric disorders, other-emotional lability (Psychiatric disorders) | 1 | 3 | 0
Psychiatric disorders - Other, Self-Injurious Behavior (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0
Psychiatric disorders - other, calmness (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders other-altered mental state (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders other-psychomotor retardation (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders, other- panic attack (Psychiatric disorders) | 0 | 0 | 1
Psychiatric disorders, other-pressured speech (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders, other-Nicotine Dependence (Psychiatric disorders) | 8 | 2 | 1
Psychiatric disorders-other (crying) (Psychiatric disorders) | 4 | 1 | 1
Restlessness (Psychiatric disorders) | 16 | 14 | 2
Somnolence (Psychiatric disorders) | 17 | 26 | 6
Suicidal ideation (Psychiatric disorders) | 0 | 3 | 0
other Sleep Disturbances (Psychiatric disorders) | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0
Renal and urinary disorders-other hematospermia (Renal and urinary disorders) | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 9 | 9 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 0
Urine output decreased (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 1
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0
Libido decreased (Reproductive system and breast disorders) | 4 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0
Reproductive system and breast disorders other - Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Reproductive system and breast disorders-other: uterine cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased Coughing (Respiratory, thoracic and mediastinal disorders) | 24 | 20 | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, mucopurulent sputum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other-Heavy Breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic, & mediastinal disorders, other-exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 37 | 34 | 18
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 15 | 9 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 3
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 17 | 13 | 6
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1 | 2
Surgical and medical Procedures - Other, Eye Surgery (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures - Other, Eye Surgery (II) (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures - Other, Eye Surgery (III) (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures - Other, exploratory endoscopy (Surgical and medical procedures) | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 2 | 0
Surgical and medical procedures - Other, tooth extraction (Surgical and medical procedures) | 1 | 2 | 0
Surgical and medical procedures - Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 0
Surgical and medical procedures - back surgery (Surgical and medical procedures) | 0 | 1 | 0
Surgical and medical procedures -other, biopsy of prostate (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures, other-removal of facial cyst (Surgical and medical procedures) | 0 | 10 | 0
Surgical and medical procedures, other-Removal of cyst (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures, other-root canal (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 8 | 3 | 0
Hypertension (Vascular disorders) | 3 | 4 | 1
Hypotension (Vascular disorders) | 1 | 2 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
Vascular disorder, other-sweating (Vascular disorders) | 3 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT00943618/Prot_SAP_000.pdf